CLINICAL TRIAL: NCT00957099
Title: A Comparison Study of Contrast Enhanced Breast CT With MRI On Known Malignancies For Detection of Multifocal/Multicentric Disease
Brief Title: Comparison Study of Breast Computed Tomography (CT) With Magnetic Resonance Imaging (MRI)
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ioannis Sechopoulos, Ph.D., Assistant Professor of Radiology and Imaging Sciences, Emory University
Other Study IDs: IRB00014357
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Imaging: Women diagnosed with breast cancer having pre-treatment MRI for spread of disease

SUMMARY:
Lay Summary

After patients are diagnosed with breast cancer, they undergo breast magnetic resonance (MR) imaging to determine if the cancer is located in more than one place in the breast. Breast MR imaging is a good option for this test because it has very high sensitivity (catches almost all breast tumors). However, breast MR is slow: it takes about two minutes to acquire one image, and is very low resolution. The points that make up the breast MR image are around 1 to 3 mm in size.

Dedicated breast computed tomography (or breast CT), a new way of imaging the breast, has been introduced in the last few years. Breast CT is an x-ray exam that uses 3D imaging to show the breast in its real three dimensional shape. Combined with the use of special chemicals called iodine contrast enhancement, breast CT can provide images of both the anatomy and the blood flow in the breast. As opposed to breast MR, breast CT is very fast. An image can be taken in 10 seconds, and has very high resolution. The points in the breast CT image are only 0.14 mm in size. The investigators propose to use breast CT instead of breast MR imaging to determine if the patient's breast cancer is located in more than one place. This is the first time anybody has proposed to use breast CT for this, so the investigators aim to test the feasibility of the idea with only 6 patients.

Since the patients will undergo breast MR as part of the standard of care, the investigators will be able to compare the breast CT images to the current standard, breast MR. This work will lay a foundation for performing this very important test before breast cancer treatment planning with a new, fast, high resolution imaging method, breast CT.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
3.1 Eligibility Criteria All subjects will be women at least 35 years of age that have been diagnosed with breast cancer and have undergone breast MR imaging for detection of multifocal/multicentric disease.

3.2 Ineligibility Criteria

* Subject does not meet any of the inclusion criteria
* Women with suspected or confirmed pregnancy
* Women who have had bilateral mastectomy
* Women who are very frail and unable to cooperate
* Women who cannot give informed consent
* Male subjects
* Women with implants

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is women who have been diagnosed with breast cancer and have undergone breast MR imaging for detection of multifocal and/or multicentric tumors before undergoing treatment.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Comparison of staging accuracy | After biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Sechopoulos, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Breast Imaging Center, Atlanta, Georgia, United States